CLINICAL TRIAL: NCT03650582
Title: Assessing the Effects of Intranasal Glucagon on Energy Balance in Humans
Brief Title: Intranasal Glucagon and Energy Balance
Acronym: INGEB
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: ING 16-5909
Record Dates: First submitted 2018-02-27; First posted 2018-08-28 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-02

CONDITIONS: Obesity
Keywords: food intake; energy expenditure; central nervous system; appetite
MeSH Terms: conditions — Obesity | interventions — Glucagon

STUDY DESIGN:
Intervention Model Description: Participants receive either glucagon or placebo as intranasal spray, in random order on 2 separate study visits, with indirect calorimetry, appetite and food intake assessment
Who Masked: Participant
Masking Description: Single-blinded study with participant blinded to treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glucagon (Experimental): Glucagon, 0.7mg, intranasal, single dose
  Interventions: Drug: Glucagon
- Placebo (Placebo Comparator): Placebo, intranasal, single dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Glucagon — Intranasal glucagon
  Arms: Glucagon
Drug: Placebo — Intranasal placebo
  Arms: Placebo

SUMMARY:
People who are overweight often find it difficult to lose weight through diet and medications because weight loss reduces the amount of energy spent by the body and increases appetite. Glucagon, when given as an injection, reduces appetite and increases the amount of energy spent by the body, even when resting. Based on studies in animals, it does so by working on the brain. However, when gives as an injection it raises blood sugar levels by acting on the liver and therefore it is not used as a weight loss drug. It has previously been shown that hormones such as glucagon, when given as a spray through the nose, can reach the brain with no major effect on the liver. Importantly it does not increase blood sugar. In this study the research team is investigating whether nasal glucagon reduces appetite and increases energy spent by the body compared to a placebo spray. If it does, it may be a potential treatment for losing weight.

DETAILED DESCRIPTION:
Resting energy expenditure, appetite and food intake is being investigated in up to 20 individuals. Participants are their own control in a single-blind, placebo-controlled, crossover design. Participants are admitted after an overnight fast and allowed to rest for 1 hour before either intranasal glucagon (0.7mg) or intranasal placebo (sterile diluent) is administered. Study visits occur 1-3 weeks apart with intranasal glucagon or placebo applied in random order. Resting energy expenditure is measured via indirect calorimetry at baseline and over 90 minutes post-spray in 10-20 minute segments. Blood samples are taken at baseline and at regular intervals post-spray to measure glucagon, glucose and other hormones/metabolites. Appetite is assessed by visual analogue scale at 90 minutes post-spray followed by provision of a buffet-style meal for ad libitum food intake measurement.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index 25- 40 kg/m2
* Hemoglobin in the normal range
* Normal fasting glucose and HbA1C
* Women of reproductive age should be on contraception (oral contraceptive pill or intra-uterine device/coil) for at least 1 month prior to and after the study.

Exclusion Criteria:

* Any history of heart disease or clinically significant, active, cardiovascular history
* Study participant with active hepatic disease (except hepatic steatosis which is frequently seen in overweight/obese individuals)
* Any current or previous history of biliary disease (including gall stones, biliary atresia and cholecystitis) or pancreatitis.
* Any current or previous history of malignancy
* Any significant active (over the past 12 months) disease of the gastrointestinal, pulmonary, neurological, renal (Cr > 1.5 mg/dL) genitourinary, hematological systems, or has severe uncontrolled treated or untreated hyper/ hypotension (sitting diastolic BP > 100 or systolic > 180 or systolic BP<100).
* Allergy to any study medication
* Pregnancy or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-06-06 (Actual); Primary Completion 2018-09-30 (Estimated); Study Completion 2018-10-30 (Estimated)

PRIMARY OUTCOMES:
Energy Expenditure | 90 minutes
  Resting energy expenditure measured by indirect calorimetry

SECONDARY OUTCOMES:
Food intake | 90 minutes
  Ad libitum food intake
Appetite | 90 minutes
  Appetite assessed by visual analogue scale ranging from 0 to 10 where 0 indicates no appetite and 10 indicates the highest appetite

CONTACTS AND LOCATIONS:
Overall Officials: Satya Dash, MD, Principal Investigator — UHN
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No